CLINICAL TRIAL: NCT05881395
Title: Assessment of Sensory Block During Labour Epidural Analgesia: a Prospective Cohort Study to Investigate the Upper and Lower Sensory Block Levels (USBL and LSBL) to Ice and Pinprick in Patients Experiencing Pain During First Stage of Labour.
Brief Title: Assessment of Sensory Block During Labour Epidural Analgesia in Patients Experiencing Pain During First Stage of Labour.
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 23-01
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Labor Pain
Keywords: epidural analgesia; sensory block; programmed intermittent epidural bolus
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with epidural analgesia experiencing pain during labor: Patients reporting pain will have their sensory block checked using ice and pinprick tests, prior to, and following and epidural top-up.

SUMMARY:
Epidural analgesia is the gold standard for pain control during labour and an essential component of delivering effective and safe epidural analgesia is the assessment of the epidural sensory block. There is significant literature on the assessment of sensory block during spinal anesthesia for cesarean section but limited studies exploring the assessment of sensory blockade in labour analgesia.

Prior studies have documented two thresholds of sensory block to both ice and pinprick: one defined as the lower sensory block level (LSBL) where the patient is able to notice a cold or sharp sensation but perceives that is not as sharp or cold as a control area and the other the upper sensory block level (USBL) where the patient perceives the cold or sharp sensation is at the same temperature or sharpness as the control area.

The goal of this study is to contribute to the standardization of the assessment of sensory block levels during labour epidural analgesia by studying patients with labour epidurals who are experiencing pain and determining the LSBL and USBL and how these change as the patients become comfortable following the administration of manual epidural top ups.

DETAILED DESCRIPTION:
The pain pathways involved in the process of labour and delivery have been well established. Nociceptive stimuli during first stage of labour are transmitted via the T10 to L1 posterior nerve root ganglia, while the nociceptive stimuli during second stage of labour are transmitted via the L1 and S2 to S4 (pudendal nerve) posterior nerve root ganglia. Although these pain pathways are well established, there is no information in the literature as to what level or depth of sensory block, assessed by current clinical practices, is required for effective labour analgesia. This information is critical for planning and safety of epidural analgesia during labour.

The investigators hypothesize that the LSBL to either cold or pinprick would be below dermatome T10 in patients receiving labour epidural analgesia during first stage of labour and who are experiencing pain. The investigators also hypothesize that upon receiving a top-up and re-establishment of effective analgesia, (a) the LSBL would be at or above dermatome T10 or (b) USBL would increase to T10 or above T10 if USBL was below T10 before receiving a top-up.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) Physical Status Classification II or III
* Patients admitted to labour and delivery unit at Mount Sinai Hospital in their first stage of labour
* Patients who have a labour epidural that has been initiated as an epidural, CSE (combined spinal epidural) or a dural puncture epidural (DPE).
* Patients who are experiencing pain, defined as Visual Numerical Rating Score of more than 1/10, despite our institution's standard epidural Programmed Intermittent Epidural Bolus maintenance regimen and request a manual epidural top-up for the first time
* Have capacity to consent to the study

Exclusion Criteria:

* Patients with a language barrier that may interfere with accurate response to sensory block assessment
* Patients with medical conditions that would compromise sensitivity to cold or pinprick assessments
* patients who sustained unintentional dural puncture, those requiring change in our standard epidural maintenance regimen or those who have had a failed epidural requiring replacement.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Patients admitted to the Labor and Delivery unit at Mount Sinai Hospital that receive epidural analgesia for labour and experience pain that is addressed by the anesthesiologist.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Lower sensory block level to ice when the patient is experiencing pain | 5 minutes
  The lower sensory block level to ice, defined as the dermatome at which there is a complete loss of cold perception. This will be checked when the patient is experiencing pain and requesting manual administration of an epidural bolus.
Upper sensory block level to ice when the patient is experiencing pain | 5 minutes
  The upper sensory block level to ice is defined as the dermatome at which there is an altered cold perception without complete sensitivity loss.This will be checked when the patient is experiencing pain and requesting manual administration of an epidural bolus.
Lower sensory block level to pinprick when the patient is experiencing pain | 5 minutes
  The lower sensory block level to pinprick, defined as the dermatome at which there is a complete loss of sharp sensation. This will be checked when the patient is experiencing pain and requesting manual administration of an epidural bolus.
Upper sensory block level to pinprick when the patient is experiencing pain | 5 minutes
  The upper sensory block level to pinprick is defined as the dermatome at which there is an altered sharp sensation without complete sensitivity loss. This will be checked when the patient is experiencing pain and requesting manual administration of an epidural bolus.

SECONDARY OUTCOMES:
Verbal Numeric Rating Score (VNRS) at the time of request of assessment by anesthesiologist | 5 minutes
  The patient will be asked to report their VNRS (0-10), where 0 is no pain and 10 is the worst pain imaginable
Verbal Numeric Rating Score (VNRS) at 10 minutes after each epidural top-up administered. | 10 minutes
  The patient will be asked to report their VNRS (0-10), where 0 is no pain and 10 is the worst pain imaginable, 10 minutes after epidural top-ups are administered.
Lower sensory block level to ice following epidural top-up | 5 minutes
  The lower sensory block level to ice, defined as the dermatome at which there is a complete loss of cold perception. This will be checked 10 minutes following each top-up or when the patient's pain is reported as 0 or 1.
Upper sensory block level to ice following epidural top-up | 5 minutes
  The upper sensory block level to ice is defined as the dermatome at which there is an altered cold perception without complete sensitivity loss. This will be checked 10 minutes following each top-up or when the patient's pain is reported as 0 or 1.
Lower sensory block level to pinprick following epidural top-up | 5 minutes
  The lower sensory block level to pinprick, defined as the dermatome at which there is a complete loss of sharp sensation. This will be checked 10 minutes following each top-up or when the patient's pain is reported as 0 or 1.
Upper sensory block level to pinprick following epidural top-up | 5 minutes
  The upper sensory block level to pinprick is defined as the dermatome at which there is an altered sharp sensation without complete sensitivity loss. This will be checked 10 minutes following each top-up or when the patient's pain is reported as 0 or 1.
Motor block score using Bromage score at the time of request of assessment by anesthesiologist | 5 minutes
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle. This will be checked when the patient is experiencing pain and requesting manual administration of an epidural bolus.
Motor block score using Bromage score following epidural top-up | 5 minutes
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle. This will be checked 10 minutes following each top-up or when the patient's pain is reported as 0 or 1.
Number of epidural top-ups required | 20 minutes
  The number of epidural top-ups documented by the anesthesiologist that were required to achieve VNRS of 0 or 1.
Type of pain: questionnaire | 20 minutes
  Patients will be asked to describe their pain as: sharp/dull/pressure.
Location of pain: questionnaire | 20 minutes
  Patients will be asked to describe the location of their pain as: abdomen/back/perineum

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kordich L, Ghiringhelli JP, George RB, Downey K, Ye XY, Carvalho J. Characterizing patterns of sensory loss during labor epidural analgesia: a prospective study of breakthrough pain. Int J Obstet Anesth. 2025 Nov;64:104753. doi: 10.1016/j.ijoa.2025.104753. Epub 2025 Aug 12. PMID 40876244